CLINICAL TRIAL: NCT01002209
Title: Postoperative Hyperbaric Oxygen Treatments to Reduce Complications in Diabetic Patients Undergoing Vascular Surgery (HODiVA) - A Double Blind, Randomized Controlled Study
Brief Title: Postoperative Hyperbaric Oxygen Treatments to Reduce Complications in Diabetic Patients Undergoing Vascular Surgery
Acronym: HODiVA
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Changes in the organisation
Sponsor: Karolinska Institutet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HODIVA
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Diabetes; Peripheral Arterial Disease; Arterial Occlusive Disease
Keywords: Diabetes; Vascular Surgery; Hyperbaric oxygen; Surgical complications; Wound complication; Randomized; Controlled
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Arterial Disease; Arterial Occlusive Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham Hyperbaric Oxygen Treatment (Sham Comparator)
  Interventions: Procedure: Sham HBO
- Hyperbaric oxygen treatment (HBO) (Experimental)
  Interventions: Procedure: Hyperbaric Oxygen treatment (HBO)

INTERVENTIONS:
Procedure: Hyperbaric Oxygen treatment (HBO) — HBO treatment will be given in a monoplace chamber and will start on first postoperative day (study day 1). The HBO group will be treated with 100% oxygen at 2.5 bar for 100 min with two 10 min airbrakes (without mask).
  HBO treatment will be given twice daily first three days (study day 1-3) and then once daily for up to three days (study day 4-6). The total number of treatments will be at least 6 and at most 9 treatments. Patients who have received at least three days HBO/placebo treatment and who have a clearly uncomplicated postoperative course will terminate HBO/placebo treatment on the day of discharge from hospital.
  Arms: Hyperbaric oxygen treatment (HBO)
Procedure: Sham HBO — HBO sham treatment will start on first postoperative day (study day 1). HBO sham treatment will be given twice daily first three days (study day 1-3) and then once daily for up to three days (study day 4-6). The total number of treatments will be at least 6 and at most 9 treatments. Patients who have received at least three days HBO sham treatments and who have a clearly uncomplicated postoperative course will terminate HBO sham treatment on the day of discharge from hospital.
  For patient blinding purposes, the sham group will breathe air and will be given a brief compression to 1.5 bar at the beginning of each treatment after which the chamber is slowly decompressed to 1.1, 1.2 , 1.3, or 1.4 bar corresponding to 0.23 ,0.25, 0.27, and 0.29 bar inspired oxygen. Two 10 min "airbrakes" will also be included.
  Arms: Sham Hyperbaric Oxygen Treatment

SUMMARY:
This trial aims to evaluate if hyperbaric oxygen treatment (HBO) given postoperatively is effective in reducing healing time and wound complications after lower extremity bypass surgery in patients with diabetes.

Hypothesis: Postoperative HBO treatment is effective in reducing complications in patients with diabetes undergoing peripheral vascular surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for inclusion if the following criteria are fulfilled
* Informed consent obtained
* Scheduled for lower extremity open vascular surgery
* Diabetes treated with insulin or oral antidiabetic medicine
* Age ≥ 18 years

Exclusion Criteria:

* Contraindications to HBO therapy
* Pregnancy (women of childbearing potential will undergo pregnancy test before inclusion)
* Patients already in HBO treatment
* Vascular reoperation
* Creatinine > 250 mmol/L
* NYHA class IV heart failure or severe cardiopulmonary disease with desaturation judged to be incompatible with safe HBO/ placebo therapy in a monoplace chamber
* Clinically significant chronic obstructive pulmonary disease.
* Acute sepsis.
* Malignancy or other serious medical condition where it is likely that the patient will significantly deteriorate or not survive within the two years of follow up.
* Simultaneous or previous (within 30 days prior to study entry participation in a clinical study using experimental drugs or devices.
* Mental condition making the subject unable to understand the concepts and risk of the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Time to complete healing of operative wounds | 7-365 days

SECONDARY OUTCOMES:
Number of wound infections at 7 days assessed by ASEPSIS score. A score over 20 will be considered as a wound infection. | 7 days (plus minus 3 days)
Number of wound infections at 30 days assessed by ASEPSIS score. A score over 20 will be considered as a wound infection. | 30 days (plus minus 3 days)
The severity of wound infection defined as by ASEPSIS score: 0-10= satisfactory healing 11-20= disturbed healing 21-30= minor wound infection 31-40= moderate wound infection >40= severe wound infection. | highest score up to 30 days (plus minus 3 days)
A combination of any wound infection and/or unhealed wounds at 30 days (combined endpoint). | 30 days (plus minus 3 days)
SF-36 score | 7, 14, 28, 365 days (plus minus 3 days)
Major amputation or death. This will be assessed as "amputation-free survival". A major amputation is defined as any ipsilateral amputation through or above the ankle. | 0-365 days
Tissue perfusion and oxygenation on dorsum of foot on operated extremity as assessed by Transcutaneous oximetry during normobaric air breathing and after 6 min normobaric 100% oxygen challenge | day 3-5, 7 and 14, 28, 365 (plus minus 3 days)
HBO complications (confinement anxiety, barotrauma, oxygen convulsions) | During HBO treatment up to day 6

CONTACTS AND LOCATIONS:
Overall Officials: Kerstin Brismar, Professor, Study Director — Karolinska Institutet; Jonas Malmstedt, MD, Principal Investigator — Karolinska Institutet; Folke G Lind, MD, PhD, Principal Investigator — Karolinska Institutet; Sergiu Catrina, MD, PhD, Principal Investigator — Karolinska Institutet; Joy Roy, MD, PhD, Principal Investigator — Karolinska Institutet; Nils Pettersson, MD, PhD, Principal Investigator — Karolinska Institutet; Bengt M Eriksson, MD, Principal Investigator — Hyperbaric Medicine, Karolinska Univ Hosp
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden